CLINICAL TRIAL: NCT06294951
Title: Functional Magnetic Resonance Imaging Findings and Symptoms in Bladder Pain Syndrome: A Descriptive Study
Brief Title: fMRI for BPS: A Descriptive Study of Findings and Symptoms
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhebin Du, Attending Physician, RenJi Hospital
Other Study IDs: IIT-2023-0225
Record Dates: First submitted 2024-02-19; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BPS group: Patients with BPS (subject to current diagnostic criteria and clinical guidelines).
  Interventions: Diagnostic Test: fMRI
- Control group: Patients with symptoms of bladder pain and evidence of current urinary tract infection.
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — The fMRI is acquired using a Siemens 3.0T MRI scanner. BOLD functional images are scanned using an echo planar imaging (EPI) sequence. The scanning parameters are: TR=2s, matrix size of 64*64, number of layers=30, layer thickness=3.75*3.75*4.5mm, and bottom-up interval scanning. A total of 540 whole brain functional images are acquired.

SUMMARY:
The goal of this observational study is to investigate the relationship between functional magnetic resonance imaging (fMRI) findings of the brain and symptom presentation in patients with bladder pain syndrome (BPS). The main questions it aims to answer are:

1. To explore the distribution characteristics of fMRI imaging and possible target lesions in the patient population.
2. To provide appropriate clues and evidence for etiological exploration and therapeutic targeting of BPS.

Participants will undergo fMRI as well as other routine laboratory tests and queries.

DETAILED DESCRIPTION:
1. Subject management

1. Recruitment Subjects are recruited from the first consultation of patients; the specific place is the urology outpatient clinic of Renji Hospital, Shanghai Jiao Tong University School of Medicine; the specific time is from the beginning of recruiting subjects until the target of recruiting subjects is reached. If the attending physician initially judged that the criteria were met, recruitment is carried out after communication with the patient and family.
2. Informed consent After the attending physician (investigator) finds patients who initially meet the enrolment criteria, he/she should give a written and verbal explanation to the subjects on the background, nature, significance, steps, benefits, risks, compensation, injury compensation, withdrawal, etc. of the study, and must obtain an informed consent form signed by each subject (or subject's legal representative). The informed consent form is dated, and the informed consent form and its copy are kept by the investigator and the subject respectively.

   The informed consent form and its copy are kept by the investigator and the subject respectively.
3. Checking the entry criteria As soon as possible after the preliminary identification of subjects, the attending physician and the investigator will jointly check the enrolment criteria, make a formal decision on recruitment or non-recruitment into the group, and notify the subjects; the reasons for non-recruitment into the group should be explained in detail and recorded.
4. Examination of medical history and records of combined medications During the initial screening and verification of the enrollment criteria, the attending physician obtains the subject's past history, current medical history, personal history, as well as comorbid medications and previous medications. If necessary, while signing the informed consent form, the patient himself/herself or under the guidance of the attending physician will declare the medical history and combined medication records.
5. Assignment of screening numbers At the time of signing the informed consent, each patient is assigned a screening number, the rules for the preparation of the screening number are specified separately, and should ensure the principles of continuity, traceability, and de-specialization.
6. Visiting One visit is conducted on the day of signing the informed consent and one visit is conducted on the day of completion of screening, and the requirements and contents of the visit are described below.

Information to be collected on the day of signing informed consent (screening period) includes: demographic data, medical history, concomitant medications and therapies, adverse events and drug abuse; examinations and assessments to be completed include: VAS, IC-Q, PUF scale, Hamilton Depression Scale (HAMD), Hamilton Anxiety Scale (HAS), and Hamilton Anxiety Scale (HAS). (HAMD), and Hamilton Anxiety Scale (HAMA). The information collected during the screening period and the assessment results will be used as the basis for enrolment. After the decision of enrolment is made, the patients will enter the assessment period, during which the information to be collected includes: demographic data, medical history, adverse events; the tests and assessments to be completed include: urine routine, urine culture, urinary ultrasound, urodynamics, fMRI, VAS, IC-Q, PUF Scale, and Hamilton Depression Scale (HAMD), Hamilton Anxiety Scale (HAMA). Hamilton Depression Scale (HAMD), Hamilton Anxiety Scale (HAMA).

2.Data Management

1. Data entry The investigator loads the data into the case report form in a timely, complete, correct and legible manner based on the subject's original observation record. The questionnaire after review and signature by the monitor should be sent to the clinical research data manager in a timely manner.

   The entry is done using the appropriate database system of two-person dual-machine entry, after which the database is compared twice, during which the monitor is notified promptly if any problems are found, and the researcher is asked to make a reply. The exchange of various questions and answers between them should be in the form of a questionnaire, which should be kept for reference.

   Content and manner of data verification and management When all the case report forms have been double-entered and checked for accuracy, a database check report will be written by the data administrator, which will include study completion (including list of dislodged subjects), inclusion/exclusion criteria check, completeness check, logical consistency check, outlier data check, time-window check, combined medication check, and adverse event check.

   At the audit meeting, the principal investigator, representatives of the sponsor, supervisors, data managers and statisticians will make a resolution on the issues raised in the subjects' signing of the informed consent form and the database checking report, write an audit report, and the database will be locked at the same time.
2. Data archiving After completing data entry and verification as required, the case report form will be filed and kept in a numbered sequence and filled in with a search catalogue, etc., for examination. Electronic data files including databases, examination procedures, analytical procedures, analytical results, code books and description documents should be classified and kept with multiple backups on different disks or recording media for proper preservation and prevention of damage. All original files should be preserved for the period within the appropriate regulations.

3. Analysis and statistical methods

According to the basic principle of Intention-to-Treat (ITT), the analyses of the main indicators should include all subjects, regardless of whether they completed the trial or not. However, subjects who did not complete the trial should be clearly indicated in the analysis for censoring; the baseline clinical characteristics of the patients and the fMRI imaging results were statistically described, and the statistical analysis process adopted for the fMRI data is as follows: fMRI data were analyzed using the SPM8 tool, which is divided into 2 levels:

1. Individual level. The brain activation of individual subjects is assessed by linearly correlating the blood oxygen level-dependent (BOLD) sequence of each voxel with a reference function, and the voxel is considered to be significantly activated when the level of the statistical parameter is greater than a certain value. The reference function is constructed by convolutional integration of pain score sequences based on standard haemodynamic models and haemodynamic response functions based on VAS and other scores obtained during the visit.
2. Between-group level. Individual level statistics for both groups were examined using t-tests and corrected t-tests, with a p-value less than the threshold value at which the voxel is considered to be significantly different between the two groups, and the p-values of the tests for all activated voxels were mapped to a standard template of structural imagery and represented using pseudo-color coding. Significantly correlated activated brain regions were eventually labelled to show the corresponding functional patterns and potential roles played in pain formation.

ELIGIBILITY:
Inclusion Criteria for BPS group:

1. Be 18 years of age or older and female;
2. Be diagnosed with BPS (persistent or recurrent pain in the bladder area accompanied by at least one other symptom, such as increased pain when the bladder is full, and frequent urination during the day and/or at night, according to the current diagnostic criteria and clinical guidelines, without any of the conditions listed in the "Exclusion Criteria" below);
3. Persistence of symptoms for more than 6 months;
4. Visual analogue scale (VAS) of pain ≥ 4;
5. O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) score of 12 or more, with pain and nocturia domain scores >2;
6. Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF) >13;
7. No history of cystoscopy within 2 years.

Exclusion Criteria for BPS group:

1. With proliferative cystoplasty or previous surgery or any pharmacological and non-pharmacological treatment for BPS;
2. Pregnant or lactating women;
3. Contraindications to MRI;
4. Average urine output less than 40 ml or more than 400 ml;
5. Haematuria (more than 1+ in urine dipstick test);
6. Evidence of current urinary tract infection at the time of recruitment;
7. Tuberculosis of the genitourinary system or cancer of the bladder or uroepithelial cancer;
8. Recurrent urinary tract infection;
9. History of hysterectomy, mid-urethral sling, pelvic organ prolapse repair, vaginal delivery or caesarean section, prostate surgery or treatment within 6 months;
10. History of neurological disease such as cerebral infarction, multiple sclerosis, or Parkinson's disease;
11. Reliance on catheterisation; including clean intermittent catheterisation or indwelling catheterisation;
12. Planned rehabilitation therapy affecting bladder function.

Inclusion Criteria for Control group:

1. Be 18 years of age or older and female;
2. With symptoms of bladder pain (defined as persistent or recurrent pain in the bladder area accompanied by at least one other symptom, such as increased pain when the bladder is full, and frequent urination during the day and/or at night) according to current diagnostic criteria and clinical guidelines;
3. Have a pain visual analogue scale (VAS) ≥ 4;
4. Evidence of a current urinary tract infection;
5. Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF) >13;
6. No history of cystoscopy within 2 years.

Exclusion Criteria for Control group:

1. With proliferative cystoplasty or previous surgery or any pharmacological and non-pharmacological treatment for BPS;
2. Pregnant or lactating women;
3. Contraindications to MRI;
4. Average urine output less than 40 ml or more than 400 ml;
5. Tuberculosis of the genitourinary system or cancer of the bladder or uroepithelial cancer;
6. History of hysterectomy, mid-urethral sling, pelvic organ prolapse repair, vaginal delivery or caesarean section, prostate surgery or treatment within 6 months;
7. History of neurological disease such as cerebral infarction, multiple sclerosis, or Parkinson's disease;
8. Dependence on catheterisation; including clean intermittent catheterisation or indwelling catheterisation;
9. Planned rehabilitation that affects bladder function.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups or cohorts will be selected from Urology clinic of Renji Hospital, Shanghai Jiao Tong University School of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
fMRI findings | 1 day (fMRI is performed once upon the recruitment of the study subject.)
  The fMRI is acquired using a Siemens 3.0T MRI scanner. BOLD functional images are scanned using an echo planar imaging (EPI) sequence. The scanning parameters are: TR=2s, matrix size of 64*64, number of layers=30, layer thickness=3.75*3.75*4.5mm, and bottom-up interval scanning. A total of 540 whole brain functional images are acquired.
  The relevant data acquired from fMRI should undergo the following pre-processing before generating findings: (1) data format conversion; (2) temporal layer correction; (3) head movement correction; (4) normalization; (5) smoothing

CONTACTS AND LOCATIONS:
Overall Officials: Zhebin Du, Dr., Principal Investigator — RenJi Hospital; Yinghui Fan, Dr., Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided